CLINICAL TRIAL: NCT00064870
Title: National Centralized Repository for Alzheimer's Disease and Related Dementias (NCRAD)
Brief Title: Alzheimer's Disease Genetics Study
Acronym: NCRAD
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Tatiana Foroud, Department Chair, Indiana University
Other Study IDs: IA0042; U24AG021886 (NIH); NIH grant U24 AG21886
Record Dates: First submitted 2003-07-14; First posted 2003-07-16 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Late Onset Alzheimer Disease; Dementia
Keywords: Alzheimer disease; Late Onset Alzheimer disease risk factor genes; Genetics; Initiative; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples, brain tissue, cell lines
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the Alzheimer's Disease Genetics Study is to identify the genes that are responsible for causing Alzheimer's Disease (AD). One of the ways in which the risk factor genes for late onset AD can be investigated is by identifying and collecting genetic material from families with multiple members diagnosed with AD or dementia.

DETAILED DESCRIPTION:
The purpose of the Alzheimer's Disease Genetics Study is to help identify the genes that may be responsible for causing Alzheimer's Disease (AD) by collecting genetic material from families with multiple members diagnosed with AD. Qualifying families will have two living blood-related individuals who have been diagnosed with or are showing symptoms of AD or dementia. Local study sites are located all over the United States, and arrangements may be made for eligible families who do not live near a participating site. The biological samples and data from these families will be made available to qualified researchers, who must sign a Materials Transfer Agreement (MTA) in order to protect the privacy rights of study participants before receiving samples and data.

ELIGIBILITY:
Inclusion Criteria:

* Two living family members diagnosed with AD or other dementia with any age of onset
* Biological samples available

  * Fresh blood, or
  * Immortalized lymphoblastic cell lines, or
  * 3-5 grams of frozen cerebral cortex; fixed samples are not accepted

Please note: this study does not include genetic counseling; because no personal identifying information such as name or date of birth is attached to samples, results of individual tests are not available to participants or family members.

Exclusion Criteria:

* Does not meet inclusion criteria
* Member of a family that was included in the National Institute of Mental Health AD Genetics Sib Pair collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Families with two or more members with Alzheimer's disease or dementia
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2002-06; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Distribute biological specimens to qualified investigators for use in their research studies. | Contact investigators annually for an update on progress and publication status.
  Investigators will analyze the samples and publish de-identified results. These publications will help to further the knowledge in the field of dementia and potentially lead to new therapies and targets for therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana M. Foroud, PhD, Principal Investigator — National Centralized Repository for Alzheimer's Disease and Related Dementias (NCRAD), Indiana University
Locations (1):
- Participants are being recruited from all over the United States, Nationwide, Indiana, United States

REFERENCES:
- See also: NCRAD: the National Centralized Repository for Alzheimer's Disease and Related Dementias — https://www.ncrad.org/